CLINICAL TRIAL: NCT00462306
Title: Incidence of Obstructive Sleep Apnea in Pregnancy
Acronym: OSA
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Cynthia Wong, Professor of Anesthesiology, Northwestern University
Other Study IDs: 0524-026
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Results first posted 2011-05-25 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Obstructive Sleep Apnea; Pregnancy
Keywords: Obstructive Sleep Apnea; Pregnancy; Berlin Questionnaire
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregnant population: The study group consisted of pregnant women, presenting to Prentice Women's Hospital of Northwestern Memorial Hospital for spontaneous labor, induction of labor, and scheduled cesarean delivery.
  Interventions: Procedure: Survey: Berlin questionnaire
- Non-Pregnant Population: The study group consisted of non-pregnant females, presenting to Northwestern Memorial Hospital for ambulatory surgery
  Interventions: Procedure: Survey: Berlin questionnaire

INTERVENTIONS:
Procedure: Survey: Berlin questionnaire — Completion of questionnaire

SUMMARY:
Obstructive sleep apnea is a condition characterized by obstruction of the upper airways and episodes of apnea and hypopnea during sleep. It is associated with significant adverse health effects. The incidence of obstructive sleep apnea in the general female population is approximately 2% but the incidence of obstructive sleep apnea in pregnancy is unknown. There is some evidence that pregnancy precipitates or at least exacerbates this condition and that there may be a relationship between intrauterine fetal growth retardation and maternal preeclampsia. In addition, there are several anesthetic implications that are concern for the patient with obstructive sleep apnea. These include: exquisite sensitivity to all central nervous system depressant drugs and the potential for upper airway obstruction or apnea with even minimal drug doses; difficult mask ventilation; difficult intubation; arterial hypoxemia; arterial hypercarbia; polycythemia; hypertension; pulmonary hypertension and cardiac failure. All of these conditions pose significant anesthetic risk for the patient, and this risk may be increased further by pregnancy.

DETAILED DESCRIPTION:
All patients presenting to the Prentice Women's Hospital's (PWH) Labor and Delivery Unit for spontaneous labor, induction of labor and scheduled cesarean delivery are routinely interviewed by a member of the anesthesia team to obtain a detailed history and physical examination and to discuss labor analgesia options. Immediately following this usual and customary preanesthetic evaluation the member of the anesthesia team performing the preanesthetic consultation (anesthesiology attending, resident physician, or nurse) used a standard verbal consent script to obtain verbal consent from the subject for study participation. Study participants were asked to complete a written validated survey, the Berlin Questionnaire, evaluating self-reported snoring and daytime sleepiness as well as basic demographic data (age, height, current weight and pregnancy weight gain). Survey completion time was 1 to 2 minutes.

The survey was available in English and Spanish. It did not contain any subject personal health information. The survey sheet remained in the labor and delivery room with the subject's usual anesthesia medical record paperwork until the patient was discharged from the unit. At the time of discharge, the infant's birthweight and APGAR scores were recorded on the survey and the survey collected.

All female patients, ages 18 - 45, presenting to the PWH Operating Room for elective gynecologic surgery, and all female patients, ages 18 - 45, presenting to the Northwestern Memorial Hospital (NMH) Ambulatory Surgery Center were interviewed by a member of the anesthesia team to obtain a routine preoperative history and physical examination and to discuss the anesthesia options. Immediately following this usual and customary preanesthetic evaluation the member of the anesthesia team performing the preanesthetic consultation (anesthesiology attending, resident physician, or certified registered nurse anesthetist) used a standard verbal consent script to obtain verbal consent from the subject for study participation. Study participants were asked to complete a written validated survey, the Berlin Questionnaire, evaluating self-reported snoring and daytime sleepiness as well as basic demographic data (age, height, and weight). The survey was available in English and Spanish. Survey completion time was 1-2 minutes. The survey did not contain any patient identifying information and was collected after completion.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Females

  1. 18 years of age and older
  2. scheduled induction of labor
  3. spontaneously laboring
  4. scheduled cesarean delivery
* Nonpregnant Females

  1. 18 years of age or older
  2. presenting to the PWH OR for gynecologic surgery
  3. presenting to the NMH Ambulatory Surgery Center for ambulatory surgery

Exclusion Criteria:

* patient refusal
* patient age > 45 years old
* inability to understand the English language
* patient presenting for an emergency procedure

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant females spontaneously laboring, scheduled for induction of labor or scheduled for a cesarean delivery, and non-pregnant females presenting for outpatient surgery between the ages of 18-45.
Sampling Method: Non-Probability Sample
Enrollment: 4577 (Actual)
Dates: Start 2005-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Wong, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Roush SF, Bell L. Obstructive sleep apnea in pregnancy. J Am Board Fam Pract. 2004 Jul-Aug;17(4):292-4. doi: 10.3122/jabfm.17.4.292. PMID 15243018
- [Background] Young T, Peppard PE, Gottlieb DJ. Epidemiology of obstructive sleep apnea: a population health perspective. Am J Respir Crit Care Med. 2002 May 1;165(9):1217-39. doi: 10.1164/rccm.2109080. PMID 11991871
- [Background] Guilleminault C, Kreutzer M, Chang JL. Pregnancy, sleep disordered breathing and treatment with nasal continuous positive airway pressure. Sleep Med. 2004 Jan;5(1):43-51. doi: 10.1016/j.sleep.2003.07.001. PMID 14725826
- [Background] Netzer NC, Stoohs RA, Netzer CM, Clark K, Strohl KP. Using the Berlin Questionnaire to identify patients at risk for the sleep apnea syndrome. Ann Intern Med. 1999 Oct 5;131(7):485-91. doi: 10.7326/0003-4819-131-7-199910050-00002. PMID 10507956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We compared Berlin Questionnaire scores between pregnant and nonpregnant females between October 2005 through September 2007. The study group consisted of pregnant women presenting to Prentice Women's Hospital and non-pregnant females (control group) presenting to Northwestern Memorial Hospital for ambulatory surgery.
Pre-assignment Details: An anesthesia team member used a standard verbal consent script to obtain verbal consent for study participation. 4074 parturients and 503 non-pregnant women completed the Berlin Questionnaire. 13 of the non-pregnant patient questionnaires were excluded due to insufficient data.
Period: Overall Study
Arm/Group | Pregnant Population | Non-Pregnant Population
Started | 4074 | 503
Completed | 4074 | 490
Not Completed | 0 | 13
Not completed — insufficient data | 0 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnant Population | Non-Pregnant Population | Total
Number analyzed (Participants) | 4074 | 503 | 4577
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4074 | 503 | 4577
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4074 | 503 | 4577
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4074 | 503 | 4577

OUTCOME MEASURES:

1. Primary Outcome: Positive Berlin Questionnaire Indicative of Sleep Disordered Breathing
Description: The Berlin Questionnaire consists of three categories designed to elicit information regarding snoring (category 1), daytime somnolence (category 2), and the presence of obesity and/or hypertension (category 3). Categories 1 and 2 are considered positive if 2 or more responses are positive category 3 is considered positive if 1 response is positive and/or the body mass index is greater than 30 kg per meter squared. A patient is considered to have a high likelihood of sleep disordered breathing if 2 or more categories are positive.
Time Frame: 1-2 minutes
Population: Pregnant Women presenting to Prentice Women's Hospital or non-pregnant women or childbearing age presenting for ambulatory surgery from 10/2005 to 9/2007 were selected randomly and asked to complete the survey.
Measure: Number; unit: participants
Groups:
- Non-Pregnant Women: Non-pregnant women undergoing a surgical procedure
Arm/Group | Pregnant Women | Non-Pregnant Women
Number analyzed (Participants) | 4074 | 503
participants | 1343 | 96
Statistical Analysis 1: Comparison: Pregnant Women vs Non-Pregnant Women; We hypothesized that the rate of positive Berlin questionnaires would be higher in pregnant women compared to age matched controls undergoing surgery; Test type: Superiority or Other; p = 0.001, Chi-squared, Corrected — 4000 parturients and 500 non-pregnant achieves 90% power to detect a difference of 3% positive Berlin Questionnaire rates between pregnant and non-pregnant women using a two sided chi squared test at a significance level of 0.05

2. Secondary Outcome: Diagnosis of Pre-eclampsia Among Subjects With Positive Berlin Questionnaires
Description: Number of subjects with obstetrician diagnosis of pregnancy induced hypertension (pre-eclampsia) among subjects with a positive compared to a negative Berlin questionnaire. The Berlin Questionnaire consists of three categories. Categories 1 and 2 are considered positive if 2 or more responses are positive category 3 is considered positive if 1 response is positive and/or the body mass index is greater than 30 kg per meter squared. A patient is considered to have a Positive Berlin Questionnaire if 2 or more categories are positive.
Time Frame: 1-2minutes
Population: Analysis per protocol
Measure: Number; unit: participants
Groups:
- Positive Berlin Questionaires: Pregnant Women with Berlin Questionnaire Responses Indicative of Sleep Disordered Breathing
- Negative Berlin Questionnaires: Pregnant Women with Results of Berlin Questionnaire not Indicative of Sleep Disordered Breathing
Arm/Group | Positive Berlin Questionaires | Negative Berlin Questionnaires
Number analyzed (Participants) | 1343 | 2731
participants | 135 | 49
Statistical Analysis 1: Comparison: Positive Berlin Questionaires vs Negative Berlin Questionnaires; Test type: Superiority or Other; p = 0.01, Chi-squared, Corrected

ADVERSE EVENTS:
Arm/Group | Pregnant Population | Non-Pregnant Population
Serious Adverse Events (participants affected / at risk) | 0/4074 | 0/503
Other Adverse Events (participants affected / at risk) | 0/4074 | 0/503

LIMITATIONS AND CAVEATS:
The Berlin questionnaire has not been validated as a screening tool in pregnancy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes